CLINICAL TRIAL: NCT01492634
Title: Clinical Investigation Plan Optimizing Fluid Status
Brief Title: Optimizing Fluid Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Maduell (Other)
Collaborators: Fresenius Medical Care Europe (Unknown)
Responsible Party: Sponsor-Investigator, Francisco Maduell, Principal Investigator; Head of Dialysis Section, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HD-IIT-01-E
Record Dates: First submitted 2011-12-07; First posted 2011-12-15 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2011-12

CONDITIONS: Hypotension During Dialysis
Keywords: bioimpedance; overhydration; dry weight
MeSH Terms: conditions — Water Intoxication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Prescription of post-dialytic weight based on BCM device — Prescription of post-dialytic weight target: On a weekly base, the patients are pre-dialytically measured by BCM (body composition monitor).
  The time average fluid overload (TAFO) determines the target range. TAFO is defined as the mean value of pre- and post-dialytic overhydration (TAFO = (OHpre+OHpost)/2). The target range is set asymmetrically around a TAFO of 0.8, from -1.0 L to +0.5, i.e. the TAFO target range will be from -0.2 L to 1.3 L.
  Prescription steps will be calculated weekly for all study patients. TAFO < -0.2 L: Increase post-dialytic weight by Cw x 0.5 kg/week, TAFO between -0.2 to 1.3 L: No action, TAFO between 1.3 to 2.8 L Decrease post-dialytic weight by Cw x 0.5 kg/week, TAFO > 2.8 L: Decrease post-dialytic weight by Cw x 1.0 kg/week.
  Other Names: BCM or Body Composition Monitor Fresenius Medical Care

SUMMARY:
Title of study: Optimizing Fluid Status

Study code: HD-IIT-01-E

Study design: Prospective open design in study centre at two locations

Applied medical device: Body Composition Monitor (BCM) for determination of fluid overload and dry weight

Aim of the study: To improve the fluid status in chronic HD patients (measured as OH (overhydration) or TAFO (time averaged fluid overload)) based on BCM measurements. Up to now, the BCM was occasionally applied in both locations of the study centre.

Study hypothesis: Regular measurement of fluid status (assessed by BCM) and display of dry weight (post-weight plan)will have significant consequences, namely a decrease of the:

* time averaged fluid overload (TAFO),
* proportion of patients with severe overhydration OH > 2.5 L,or OH/ECW > 15 %)
* proportion of dehydrated patients (OH < -1.0 L, or OH < -7 %),
* mean overhydration,
* variance of overhydration,
* time outside the reference range (-1.0L < OH < 2.5L).

Devices used in this study: Dialysis machine 5008 equipped with Blood Pressure Monitor BPM, Blood Volume Monitor BVM, Blood Temperature Monitor BTM, and Online Clearance Monitor OCM ; Body Composition Monitor BCM ; Data management software / database system NephroLink Disposables used in this study: BVM blood lines and BCM electrodes

Patients: 60 patients

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal failure stage V
* Treatment thrice weekly with HD or on-line HDF for at least 6 months prior to inclusion
* Ability to understand the nature and requirements of the study
* Age: at least 18 years
* Signed informed consent.

Exclusion Criteria:

* Interventional clinical study during the preceding 30 days or previous participation in the same study
* Acute or chronic infection (HIV, Hepatitis B or C, ...)
* Severe disease (malignant tumour, tuberculosis ...)
* Usually single needle HD
* Problems with shunt or high recirculation,
* Severe intra-dialytic blood pressure instability in the last month
* Instable angina pectoris
* Major amputation at arm or leg, or a pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
intra-individual difference in TAFO between study start and study end | 3 months

SECONDARY OUTCOMES:
Comparison between start and end of treatment will be performed for Pre-dialytic overhydration (OH) | 3 months
Comparison between start and end of treatment will be performed for number of patients in target range (TAFO from -0.2 L to 1.3 L) | 3 months
SF 36 total score and sub-scores as calculated according to official guidelines, | 3 months
BNP | 3 months
Blood pressure | 3 months
laboratory parameters (sodium, calcium, potassium, chloride, haematocrit, haemoglobin, albumin, total protein, urea, creatinine, mean corpuscular volume, C-reactive protein, transferrin saturation, ferritin). | 3 months
Change from Baseline in Medication at 12 weeks (erythropoetin, iron, blood pressure medication) | 3 months
Change from baseline in intra-dialytic events (hypotension, cramps) | 3 months
Change from baseline in Residual Renal Function | 3 months
  Baseline Residual renal function, measured as Kt/V residual, wil be compared with the Residual renal function at the end of 12 weeks.
Hospitalisation | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dialysis Units, Hospital Clínic, Barcelona, Barcelona, Spain

REFERENCES:
- [Result] Moissl U, Arias-Guillen M, Wabel P, Fontsere N, Carrera M, Campistol JM, Maduell F. Bioimpedance-guided fluid management in hemodialysis patients. Clin J Am Soc Nephrol. 2013 Sep;8(9):1575-82. doi: 10.2215/CJN.12411212. Epub 2013 Aug 15. PMID 23949235